CLINICAL TRIAL: NCT01840527
Title: Exploring the Utility of a Novel BRAF Test in Patients With Melanoma
Brief Title: Utility of Novel BRAF Test for Melanoma
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Ryan J Sullivan, Principal Investigator, Massachusetts General Hospital
Other Study IDs: 12-488; 1UH2CA207355 (NIH)
Record Dates: First submitted 2013-04-23; First posted 2013-04-25 (Estimated); Results first posted 2024-09-04 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-08

CONDITIONS: Melanoma
Keywords: Biomarker; BRAF; blood-based
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood lymphocytes (PBLs); Plasma; Tumor Tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Advanced Melanoma: For patients in the advanced melanoma cohort, a one-time blood sample will be obtained prior to the commencement of systemic therapy at a time when standard-of-care blood will be drawn. While it is ideal to obtain samples prior to any systemic therapy, participants who have previously received therapy, have progressed, and are in need of additional therapy will be considered suitable for participation. Participants with known BRAF mutation (determined by standard of care tissue testing) will undergo blood draws every 4 weeks (+/- 1 week) and at the time of disease progression.
- Stage II/III Melanoma: For patients in the high-risk stage II/III cohort, a blood draw will be performed 4-8 weeks after the completion of surgical management at the time of standard of care blood work. In participants who sign informed consent prior to definite surgical management, a pre-operative blood draw may be obtained at the time that standard of care pre-op blood work is performed. Blood samples will then be obtained every three months following the initiation of either adjuvant therapy or routine, close follow-up for up to two years.

SUMMARY:
This primary purpose of this study is to obtain blood samples from participants with both early and later stages of melanoma (Stage II/III and Stage IV). The researchers hope to better understand an abnormal protein found in many melanoma tumors called the BRAFV600 mutation.

There will be two separate cohorts (groups) of participants on this study. You will be placed in one of the Groups.

Group 1-For participants with advanced melanoma: Your existing tumor tissue sample will be compared to the blood samples given in order to further analyze and to understand the BRAFV600E gene mutation.

Group 2-For participants with stage II/III melanoma: Following surgery, blood samples will be collected and analyzed.

Understanding the BRAFV600E gene mutation in melanoma will help the researchers better understand the disease, and help plan treatment options for people with melanoma of all stages in the future.

DETAILED DESCRIPTION:
There will be no extra clinic visits for this study. These research blood samples will be drawn at the same time as your regularly scheduled blood draws that are part of standard care for melanoma.

About 2 to 4 teaspoons of blood will be drawn for each research sample.

Depending on which group you are in, you will have either a one time blood draw or ongoing blood work for 1-2 years.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven advanced (unresectable stage IIIC or stage IV)or high risk (stage II or stage III) malignant melanoma

Exclusion Criteria:

* History of a different malignancy except for the following circumstances: disease-free for at least 2 years and deemed by the investigator to be at low risk for recurrence; or non-metastatic prostate cancer, cervical cancer in situ and basal cell or squamous cell carcinoma
* Known history of a different BRAF mutant malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients being treated at Massachusetts General Hospital, Dana-Farber Cancer Institute and Beth Isreal Deaconess Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2017-03-29 (Actual); Study Completion 2022-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Sullivan, MD, Principal Investigator — Massachusetts General Hospital
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Advanced Melanoma | Stage II/III Melanoma
Started | 110 | 110
Completed | 110 | 110
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Advanced Melanoma | Stage II/III Melanoma | Total
Number analyzed (Participants) | 110 | 110 | 220
Age, Continuous [Mean (Full Range); unit: years] | 59.8 [22 to 85] | 59.7 [22 to 91] | 59.7 [22 to 91]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 32 | 65
  Male | 77 | 78 | 155
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 101 | 101 | 202
  Unknown or Not Reported | 9 | 8 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 105 | 105 | 210
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 3 | 4 | 7
Region of Enrollment [Number; unit: participants]
  United States | 110 | 110 | 220

OUTCOME MEASURES:

1. Primary Outcome: Determine Sensitivity of Blood-Based Assay
Description: The specificity and sensitivity of the blood-based assay will be determined vis-à-vis tissue-based BRAF analysis in patients with advanced and high-risk melanoma in order to provide BRAF-directed therapy when indicated. The sensitivity of an assay is expressed as the probability (as a percentage) that a sample tests positive for BRAF mutation given that the participant has BRAF mutation; it is used to assess the risk of false negative results. A percentage greater than 50% indicates that the test is a better predictor of sample diagnosis than random chance.
Time Frame: 2 years
Population: The study's primary outcome was not reached because the assay has not been successfully developed so no collected samples could be analyzed. More sensitive ctDNA approaches have made their way into commercial use including bespoke assays during the course of this study. The value of a highly-sensitive BRAF specific assay seemed less useful, and given the past troubles developing the current assay approach, the study team decided to apply the philanthropic funds to other projects.
Arm/Group | Advanced Melanoma | Stage II/III Melanoma
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Determine Specificity of Blood-Based Assay
Description: The specificity and sensitivity of the blood-based assay will be determined vis-à-vis tissue-based BRAF analysis in patients with advanced and high-risk melanoma in order to provide BRAF-directed therapy when indicated. The specificity of an assay is expressed as the probability (as a percentage) that a test returns a negative result for BRAF mutation given that the that participant does not BRAF mutation; it is used to assess the risk of false positive results. A percentage greater than 50% indicates that the test is a better predictor of sample diagnosis than random chance.
Time Frame: 2 years
Population: as for outcome 1
Arm/Group | Advanced Melanoma | Stage II/III Melanoma
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Explore Pharmacodynamic Effects of MAPK Pathway Inhibitors
Description: To explore the pharmacodynamic effects of MAPK pathway inhibitors (including selective BRAF inhibitors, MEK inhibitors, and ERK inhibitors) utilizing pre-and on-treatment peripheral blood BRAFV600E mutational testing in participants with advanced melanoma.
Time Frame: 2 years
Population: as for outcome 1
Arm/Group | Advanced Melanoma | Stage II/III Melanoma
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Define Prognostic Value of Peripheral Blood BRAFV600 Testing in Melanoma
Description: To define the prognostic value of peripheral blood BRAFV600 mutational testing in participants with Stage II/III melanoma
Time Frame: 2 years
Population: as for outcome 1
Arm/Group | Advanced Melanoma | Stage II/III Melanoma
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: up to 2 years
Arm/Group | Advanced Melanoma | Stage II/III Melanoma
All-Cause Mortality (participants affected / at risk) | 68/110 | 40/110
Serious Adverse Events (participants affected / at risk) | 0/110 | 0/110
Other Adverse Events (participants affected / at risk) | 0/110 | 0/110

LIMITATIONS AND CAVEATS:
The study's primary outcome was not reached because the assay has not been successfully developed so no collected samples could be analyzed. More sensitive ctDNA approaches have made their way into commercial use including bespoke assays during the course of this study. The value of a highly-sensitive BRAF specific assay seemed less useful, and given the past troubles developing the current assay approach, the study team decided to apply the philanthropic funds to other projects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-21): https://cdn.clinicaltrials.gov/large-docs/27/NCT01840527/Prot_SAP_000.pdf